CLINICAL TRIAL: NCT00895557
Title: Assessing the Impact of Varenicline on Brain-Behavior Vulnerability in Cocaine Dependence
Brief Title: Assessing the Impact of Varenicline on Brain-Behavior Vulnerability
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study never started, no funding.
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 807134; 1P50DA012756 (NIH); Supplement (Other Grant/Funding Number: P50-DA012756); DPMC (Other: NIDA)
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Varenicline and the Blunting of Cocaine Cues
Keywords: varenicline; cocaine; brain imaging
MeSH Terms: interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- chantix (Active Comparator)
  Interventions: Drug: chantix

INTERVENTIONS:
Drug: chantix — .5 mg once a day 1 to 3, .5 mg twice a day on days 4 to 7, 1 mg from day 8 to end of treatment
  Other Names: varenicline

SUMMARY:
Our proposal will enable us to study cocaine patients to determine whether varenicline can weaken brain arousal to drug cues in an fMRI imaging setting, which is what we theorize. This supplement supports a pilot imaging study in cocaine dependence. It will evaluate the impact of varenicline on the brain response to ultra-brief drug and comparison cues in an event-related fMRI paradigm. This is a pilot study.

We will additionally examine the impact of varenicline on addiction-relevant behavioral probes of impulsivity, inhibition, attentional and affective bias. The proposed study will provide the first brain-behavioral probes of varenicline's cocaine-relevant actions in humans, and will provide the critical scientific rationale to move the agent into future collaborative clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy male substance abuse subjects age 18-55.

Exclusion Criteria:

* 1) Participation in clinical trial and receipt of investigational drug(s) during previous 60 days 2) Clinically significant cardiovascular, hematologic, hepatic, renal, neurological or endocrinological abnormalities 3) History of serious head trauma or injury causing loss of consciousness that lasted more than 3 minutes. 4) Presence of magnetically active prosthetics, plates, pins, broken needles, permanent retainer, bullets, etc. in subject's body (unless a radiologist confirms that its presence is unproblematic). A x-ray may be obtained to determine eligibility. 5) Claustrophobia or other medical condition disabling subject from lying in the MRI for approximately 60 minute

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether varenicline, as compared to placebo, can blunt the limbic activation (e.g., amygdala, ventral striatum/ventral pallidum, etc.) by ultra-brief cocaine cues using fast event-related fMRI. | End of study

SECONDARY OUTCOMES:
Varenicline (vs. placebo) may reduce positive affective bias to drug (cocaine) cues. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rose Childress, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania, United States